CLINICAL TRIAL: NCT00971880
Title: Blood Transfusions in Thalassemia Patients, Complications and Adverse Effects.
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0039-09-EMC
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Thalassemia; Sickle Cell Anemia
Keywords: Blood transfusions; Adverse events; Hepatitis C; HIV
MeSH Terms: conditions — Thalassemia; Anemia, Sickle Cell; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving blood transfusions: All the patients with blood disorders that require blood transfusions
  Interventions: Other: Clinical medical record summary

INTERVENTIONS:
Other: Clinical medical record summary — Summary of immediate and late adverse effects of blood transfusions

SUMMARY:
Patients suffering from Thalassemia or another hemoglobinopathies required regular blood transfusions. The complications and adverse effects of blood transfusions can be classified as immediate and late. Among the immediate effects the most common are allergic reactions and fever, besides congestive heart failure in patients with cardiomyopathy. The late effects are mostly related to blood transmitted infections like HIV or Hepatitis C infections.

The purpose of this study is to summarize the data of those complications in a cohort of 100 patients receiving regular blood transfusion.

DETAILED DESCRIPTION:
About 100 patients aged several months to 50 years are treated in the Pediatric Hematology Unit, most of those patients receive blood transfusions monthly. The adverse reactions were routinely recorded during each transfusion. All the patients were also screened annually for the incidence of blood transmitted infections principally HIV and Hepatitis C. All those records will be systematically screened and all the immediate or late adverse reactions and complications related to blood transfusions will be summarized.

A second goal of this study will be to control the staff strictness related to the ministry of health protocol dealing to blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving blood transfusions due to chronic hematologic disorders

Exclusion Criteria:

* Not applicable

Ages: 1 Month to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients receiving blood transfusions due to chronic hematologic disorders
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Hematology Unit and Pediatric Dpt B - HaEmek Medical Center, Afula, Israel